CLINICAL TRIAL: NCT02730546
Title: Phase 1b/2 Clinical Trial of Neoadjuvant Pembrolizumab Plus Concurrent Chemoradiotherapy With Weekly Carboplatin and Paclitaxel in Adult Patients With Resectable, Locally Advanced Adenocarcinoma of the Gastroesophageal Junction or Gastric Cardia
Brief Title: Pembrolizumab, Combination Chemotherapy, and Radiation Therapy Before Surgery in Treating Adult Patients With Locally Advanced Gastroesophageal Junction or Gastric Cardia Cancer That Can Be Removed by Surgery
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC1541; NCI-2016-00508 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 15-005311 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2016-04-01; First posted 2016-04-06 (Estimated); Results first posted 2022-08-25 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2024-04

CONDITIONS: Gastric Cardia Adenocarcinoma; Gastroesophageal Junction Adenocarcinoma; Stage IB Gastric Cancer AJCC v7; Stage II Gastric Cancer AJCC v7; Stage IIA Gastric Cancer AJCC v7; Stage IIB Gastric Cancer AJCC v7; Stage IIIA Gastric Cancer AJCC v7; Stage IIIB Gastric Cancer AJCC v7
MeSH Terms: conditions — Stomach Neoplasms | interventions — Carboplatin; Fluorouracil; dehydroftorafur; Leucovorin; Oxaliplatin; Paclitaxel; Taxes; pembrolizumab; Magnetic Resonance Spectroscopy; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (pembrolizumab, chemotherapy, radiation, surgery) (Experimental): See Detailed Description
  Interventions: Drug: Carboplatin; Procedure: Computed Tomography; Drug: Fluorouracil; Other: Laboratory Biomarker Analysis; Drug: Leucovorin Calcium; Drug: Oxaliplatin; Drug: Paclitaxel; Biological: Pembrolizumab; Procedure: Positron Emission Tomography; Radiation: Radiation Therapy; Procedure: Therapeutic Conventional Surgery

INTERVENTIONS:
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computerized Axial Tomography; computerized tomography; CT; CT SCAN; tomography
Drug: Fluorouracil — Given IV
  Other Names: 5-Fluoro-2,4(1H, 3H)-pyrimidinedione; 5-Fluorouracil; 5-Fluracil; 5-FU; AccuSite; Carac; Fluoro Uracil; Fluouracil; Flurablastin; Fluracedyl; Fluracil; Fluril; Fluroblastin; Ribofluor; Ro 2-9757; Ro-2-9757
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Leucovorin Calcium — Given IV
  Other Names: Adinepar; Calcifolin; Calcium (6S)-Folinate; Calcium Folinate; Calcium Leucovorin; Calfolex; Calinat; Cehafolin; Citofolin; Citrec; citrovorum factor; Cromatonbic Folinico; Dalisol; Disintox; Divical; Ecofol; Emovis; Factor, Citrovorum; Flynoken A; Folaren; Folaxin; FOLI-cell; Foliben; Folidan; Folidar; Folinac; Folinate Calcium; folinic acid; Folinic Acid Calcium Salt Pentahydrate; Folinoral; Folinvit; Foliplus; Folix; Imo; Lederfolat; Lederfolin; Leucosar; leucovorin; Rescufolin; Rescuvolin; Tonofolin; Wellcovorin
Drug: Oxaliplatin — Given IV
  Other Names: 1-OHP; Ai Heng; Aiheng; Dacotin; Dacplat; Diaminocyclohexane Oxalatoplatinum; Eloxatin; Eloxatine; JM-83; Oxalatoplatin; Oxalatoplatinum; RP 54780; RP-54780; SR-96669
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475
Procedure: Positron Emission Tomography — Undergo PET scan
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging
Radiation: Radiation Therapy — Undergo radiation therapy
  Other Names: Cancer Radiotherapy; Irradiate; Irradiated; irradiation; RADIATION; Radiotherapeutics; radiotherapy; RT; Therapy, Radiation
Procedure: Therapeutic Conventional Surgery — Undergo curative-intent surgery

SUMMARY:
This phase Ib/II trial studies the side effects and best way to give pembrolizumab with combination chemotherapy and radiation therapy before surgery and to see how well it works in treating adult patients with gastroesophageal junction or gastric cardia cancer that has spread from where it started to nearby tissue and can be removed by surgery. Monoclonal antibodies, such as pembrolizumab, may block tumor growth in different ways by targeting certain cells. Drugs used in chemotherapy work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Radiation therapy uses high energy x-rays to kill tumor cells and shrink tumors. Giving pembrolizumab, combination chemotherapy, and radiation therapy before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety and tolerability of pembrolizumab when combined with radiotherapy plus carboplatin and paclitaxel in locally advanced gastroesophageal junction (GEJ)/cardia adenocarcinoma. (Phase Ib) II. To evaluate the pathological complete response (pathCR) rate of pembrolizumab when combined with radiotherapy plus carboplatin and paclitaxel in locally advanced GEJ/cardia adenocarcinoma. (Phase II)

SECONDARY OBJECTIVES:

I. To determine progression-free survival (PFS), determine time to relapse (TTR), disease-free survival (DFS), R0 rate, and overall survival (OS) of pembrolizumab when combined with radiotherapy plus carboplatin and paclitaxel.

TRANSLATIONAL RESEARCH OBJECTIVES:

I. To identify tissue and/or circulating biomarkers that are associated with pathCR, DFS, and other clinical outcomes in patients with locally advanced GEJ/cardia adenocarcinoma treated with neoadjuvant pembrolizumab-based therapy.

II. To determine differences in pre-treatment vs post-treatment tissue expression of immune markers, including PDL1 and tumor infiltrating lymphocytes (CD8+, FOXP3+ Tregs, CD45RO, granzyme B), in patients treated with neoadjuvant pembrolizumab-based therapy.

III. To identify immune markers in pretreatment tissues that correlate with pathCR and long-term outcome in patients treated with neoadjuvant pembrolizumab-based therapy.

IV. To explore whether an EBV-associated tumor molecular profile89 is associated with pathCR and long-term outcome in patients treated with neoadjuvant pembrolizumab-based therapy.

V. To explore whether a microsatellite-unstable (MSI) tumor molecular profile89 is associated with pathCR and long-term outcome in patients treated with neoadjuvant pembrolizumab-based therapy.

OUTLINE:

NEOADJUVANT TREATMENT: Patients receive pembrolizumab intravenously (IV) over 30 minutes on days -7, 15, and 36 and carboplatin IV and paclitaxel IV over 1-96 hours on days 1, 8, 15, 22 and 29. Patients also undergo radiation therapy once daily (QD) 5 days per week for 4 weeks and 3 days (23 fractions).

Patients with progressive disease receive pembrolizumab IV over 30 minutes, paclitaxel IV over 1-96 hours, and carboplatin IV on day 1. Treatment repeats every 21 days for 2-4 courses in the absence of disease progression or unacceptable toxicity.

NEOADJUVANT TREATMENT (RE-INITIATED): Patients receive pembrolizumab IV over 30 minutes on days 1 and 22 and oxaliplatin IV over 2-6 hours, leucovorin calcium IV over 15 minutes to 2 hours, and fluorouracil IV over 46-48 hours on days 1, 15, and 29. Treatment repeats every 21 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.

Patients with progressive disease receive pembrolizumab IV over 30 minutes on days 1 and 22, oxaliplatin IV over 2-6 hours, leucovorin calcium over 15 minutes to 2 hours, and fluorouracil IV over 46-48 hours on days 1, 15, and 29. Treatment repeats every 41 days (6 weeks) for 1-3 courses in the absence of disease progression or unacceptable toxicity.

SURGERY: Within 5-8 weeks after completion of radiation therapy or 3-6 weeks after completion of chemotherapy for patients receiving chemotherapy alone, patients undergo curative-intent surgery.

ADJUVANT TREATMENT: Patients receive pembrolizumab IV over 30 minutes every 21 days. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days, every 3 months for 1 year, every 4 months for 1 year, and then every 6 months for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma involving the gastroesophageal junction or gastric cardia
* Central pathology review to determine evaluability of archived esophagogastroduodenoscopy (EGD)/biopsy sample

  * NOTE: If archived sample was collected > 8 weeks prior to pre-registration (reg), is not available in a timely manner, or was collected outside of Mayo Clinic and considered unevaluable, then baseline EGD with primary tumor biopsy at Mayo Clinic must be performed unless clinically contraindicated; patient is allowed to enroll regardless of whether this Mayo Clinic tissue sample is evaluable; (Only 1 EGD with primary tumor biopsy performed at Mayo Clinic =< 8 weeks prior to pre-reg is required)
  * NOTE: For both archival or newly obtained tissue, only biopsies are adequate (fine needle aspiration [FNA] is not adequate)
* Willing to provide mandatory tissue samples for research purposes
* Baseline imaging with an fludeoxyglucose (FDG)-positron emission tomography (PET) scan negative for distant metastatic disease must be obtained =< 28 days prior to registration
* Surgically resectable (T2N0, T3N0, Tany with node positivity, M0), as determined by endoscopic ultrasound (EUS) and the following minimum diagnostic work-up:

  * Whole-body PET/computed tomography (CT) (PET/CT of skull base to mid-thigh is acceptable)
  * EUS =< 21 days prior to registration
  * NOTE: Patients may have regional adenopathy including para-esophageal, gastric, gastrohepatic and celiac nodes; if celiac adenopathy is present, it must be < 2 cm
  * NOTE: If patient unable to have PET/CT then CT chest/abdomen/pelvis with contrast (preferred) or MRI chest/abdomen/pelvis with contrast
* Surgical consultation at enrolling site to confirm that patient will be able to undergo curative resection after completion of chemoradiation =< 56 days prior to registration

  * Tumor is amenable to standard resection and reconstruction
* Radiation oncology consultation at enrolling site to confirm that disease can be encompassed in a radiotherapy field =< 56 days prior to registration

  * NOTE: Radiotherapy quality assurance rapid review must be performed before the first fraction of radiation therapy (RT) is administered; if RT constraints cannot be met, the patient will be removed from the protocol prior to treatment
* Consultation with a medical oncologist at enrolling site =< 56 days prior to registration, with determination that treatment with neoadjuvant chemoradiotherapy with weekly carboplatin and paclitaxel is considered acceptable
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Adequate oral intake and nutritional status without current or likely need for enteral or parenteral feeding during chemoradiation or the preoperative period
* Pre-treatment pulmonary function tests (PFTs), collected =< 90 days prior to enrollment, must show forced expiratory volume in one second (FEV1) > 60% of predicted
* Adequate organ function =< 21 days prior to registration:

  * Aspartate transaminase (AST) level =< 2.5 x upper limit of normal (ULN) and alanine transaminase (ALT) =< 3 x upper limit of normal (ULN)
  * Total bilirubin level of =< 1.5 x ULN
  * Creatinine level =< 1.2 x ULN or creatinine clearance > 60 mL/min/1.73 m^2 for patients with creatinine levels above or below the institutional normal
  * Hemoglobin (Hgb) >= 9 g/dl without transfusion or epoetin dependency (=< 7 days prior to assessment)
  * Absolute neutrophil count >= 1.5 x 10^9/L
  * Platelets >= 100 x 10^9/L
  * Albumin >= 2.5 g/dl
* Female patients of childbearing potential must be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication

  * NOTE: Patients of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year
* Female patients of childbearing potential must have a negative urine or serum pregnancy test =< 7 days prior to registration

  * NOTE: If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Male patients must agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy

  * NOTE: Abstinence is acceptable if this is the established and preferred method of contraception for the subject
* Provide signed written informed consent
* Willing to return to enrolling institution for follow-up
* Willing to provide mandatory tissue and blood samples for research purposes

  * NOTE: Patients must be willing to provide at the time surgical resection; for patients who do not undergo surgery, any on-study tumor biopsy obtained for clinical purposes subsequent to the baseline biopsy must also be available for analysis

Exclusion Criteria:

* Tumor characteristics - any of the following are excluded:

  * Evidence of distant metastases
  * Tumors whose location is restricted to the tubular esophagus (i.e., without involvement of the GEJ or cardia)
  * Tumors whose proximal end are at the level of the carina or higher
  * Invasion of the tracheobronchial tree or presence of tracheoesophageal fistula
  * Palpable supraclavicular nodes, biopsy-proven involvement of supraclavicular nodes, or radiographically involved supraclavicular nodes (> 1.5 cm in greatest dimension)
  * T1N0M0, T4Nany, or in situ carcinoma
  * Tumor must not extend 5 or more cm into the stomach
* Received prior treatment or receiving current treatment for this malignancy
* Prior radiation to chest or abdomen, or to > 30% of the marrow cavity
* Inadequate caloric or fluid intake whereby there is a current or likely future need for enteral or parenteral feeding during chemoradiation or the preoperative period
* Major surgery =< 4 weeks prior to registration
* Active autoimmune disorders, including patients known to be human immunodeficiency virus (HIV) positive, or those requiring chronic steroid administration (excluding inhaled steroids)
* Uncontrolled diabetes (i.e., will interfere with the performance of the FDG PET/CT scans)
* Prior allergic reactions to drugs containing Cremophor, such as teniposide or cyclosporine, or study drugs involved in this protocol, or to a monoclonal antibody or prior hypersensitivity to platinum-containing agents
* Heart conditions - any of the following:

  * Any atrial fibrillation =< 3 months prior to registration
  * Unstable angina =< 12 months prior to registration
  * Prior symptomatic congestive heart failure
  * Documented myocardial infarction =< 6 months prior to registration (pretreatment electrocardiogram [ECG] evidence of infarct only will not exclude patients)
  * Prior significant ventricular arrhythmia requiring medication
  * Prior 2nd or 3rd degree heart block or other types of clinically significant conduction delay =< 6 months prior to registration
  * Clinically significant pericardial disease (including pericardial effusion, pericarditis) or cardiac valvular disease =< 12 months prior to registration
  * NOTE: As part of history and physical, all patients must be assessed for signs or symptoms of cardiac disease, or for prior history of cardiac disease; these conditions include but are not limited to diseases related to cardiac valves, pericardium, myocardium, atrioventricular delays or arrhythmias; it is strongly recommended that signs or symptoms of potentially clinically significant disease be evaluated with comprehensive cardiac echo
* Prior pancreatitis that was symptomatic or required medical intervention =< 6 months prior to registration (known toxicity of pembrolizumab)
* Prior enteritis that was symptomatic or required medical intervention =< 6 months prior to registration (known toxicity of pembrolizumab)
* Uncontrolled hyper/hypothyroidism or hyper/hypocorticism =< 6 months prior to registration (known toxicity of pembrolizumab)
* Pulmonary conditions - any of the following:

  * Respiratory condition that required any oxygen supplementation =< 6 months prior to registration
  * Prior or current pneumonitis
  * Clinically significant pulmonary hypertension =< 12 months prior to registration
  * Lung infection requiring treatment =< 3 months prior to registration
  * Pulmonary embolism requiring treatment =< 6 months prior to registration
  * Pleural effusion requiring drainage =< 12 months prior to registration
* Prior fistula within thorax, including bronchoalveolar or esophageal
* Body mass index (BMI) >= 35 mg/m^2 =< 56 days prior to registration
* Pre-existing motor or sensory neurotoxicity greater than Common Terminology Criteria for Adverse Events (CTCAE) grade 1
* Acute bacterial, viral, or fungal infection requiring treatment at the time of registration
* Active infection or other serious underlying medical condition which would impair the ability of the patient to receive the planned treatment
* Uncontrolled intercurrent illness including, but not limited to, psychiatric illness/social situations, or other co-morbid systemic illnesses or severe concurrent diseases which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Prior malignancy =< 5 years prior to registration (except non-melanotic skin cancer or carcinoma-in-situ of the cervix) (must be disease free for a minimum of 5 years); if there is a history of prior malignancy, patient must not be receiving other specific treatment (other than hormonal therapy) for cancer
* Dementia or altered mental status that would prohibit the understanding and giving of informed consent
* Any of the following because this study involves an agent where the genotoxic, mutagenic and teratogenic effects are unknown:

  * Pregnant or breastfeeding
  * Patient of childbearing potential who is unwilling to employ adequate contraception
* Received live vaccine =< 30 days prior to registration

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2016-06-24 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2023-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harry H. Yoon, M.D., Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic Hospital, Phoenix, Arizona
  - Mayo Clinic, Rochester, Minnesota

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Pembrolizumab, Chemotherapy, Radiation, Surgery): See Detailed Description>
  > Carboplatin: Given IV>
  > Computed Tomography: Undergo CT scan>
  > Fluorouracil: Given IV>
  > Laboratory Biomarker Analysis: Correlative studies>
  > Leucovorin Calcium: Given IV>
  > Oxaliplatin: Given IV>
  > Paclitaxel: Given IV>
  > Pembrolizumab: Given IV>
  > Positron Emission Tomography: Undergo PET scan>
  > Radiation Therapy: Undergo radiation therapy>
  > Therapeutic Conventional Surgery: Undergo curative-intent surgery
Period: Overall Study
Arm/Group | Treatment (Pembrolizumab, Chemotherapy, Radiation, Surgery)
Started | 31
Completed | 31
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Pembrolizumab, Chemotherapy, Radiation, Surgery)
Number analyzed (Participants) | 31
Age, Continuous [Median (Full Range); unit: years] | 62 [44 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 31
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 31
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 31
Tumor Location [Count of Participants; unit: Participants]
  Gastroesophageal junction | 29
  Gastric cardia | 2
Histologic Grade (differentiation) [Count of Participants; unit: Participants]
  G2 (moderately differentiated) | 18
  G3 (poorly differentiated) | 12
  GX (grade cannot be assessed) | 1
Clinical Tumor Stage [Count of Participants; unit: Participants] — Size and extent of the primary tumor; higher number tumor stage indicates a larger and more invasive tumor.
  T0 No evidence of primary tumor T1 Tumor invades the lamina propria, muscularis mucosae, or submucosa T2 Tumor invades the muscularis propria T3 Tumor invades adventitia T4 Tumor invades adjacent structures
  Participants
    T2 | 2
    T3 | 29
Clinical Nodal Stage [Count of Participants; unit: Participants] — Regional lymph node involvement of the tumor; a higher number indicates more involvement of regional lymph nodes.
  N0 No regional lymph node metastasis N1 Metastasis in 1-2 regional lymph nodes N2 Metastasis in 3-6 regional lymph nodes N3 Metastasis in 7 or more regional lymph nodes
  Participants
    N0 | 4
    N1 | 13
    N2 | 12
    N3 | 2
Signet Ring Cell Histology [Count of Participants; unit: Participants] — Having a signet ring cell histology is associated worse disease outcomes.
  Participants
    Yes | 6
    No | 25
PD-L1 Combined Positive Score (CPS) [Count of Participants; unit: Participants] — Higher PD-L1 CPS corresponds to a greater likelihood of responding effectively to anti-PD-1 therapy
  Participants
    <1 | 11
    1-9 | 11
    ≥10 | 8
    Unknown | 1

OUTCOME MEASURES:

1. Primary Outcome: Pathological Complete Response (PathCR) Rate
Description: Defined as number of patients with pathologic complete responses (pCR) divided by total evaluable patients. pCR is defined as no recognized cancer and margins free of tumor as found by the pathologist following resection of the esophageal specimen and accompanying lymph nodes.
Time Frame: Up to 3 years
Measure: Number (95% Confidence Interval); unit: percentage of patients
Groups:
- Treatment (Pembrolizumab, Chemotherapy, Radiation, Surgery): See Detailed Description >
  > Carboplatin: Given IV
  >
  > Computed Tomography: Undergo CT scan
  >
  > Fluorouracil: Given IV
  >
  > Laboratory Biomarker Analysis: Correlative studies
  >
  > Leucovorin Calcium: Given IV
  >
  > Oxaliplatin: Given IV
  >
  > Paclitaxel: Given IV
  >
  > Pembrolizumab: Given IV
  >
  > Positron Emission Tomography: Undergo PET scan
  >
  > Radiation Therapy: Undergo radiation therapy
  >
  > Therapeutic Conventional Surgery: Undergo curative-intent surgery
Arm/Group | Treatment (Pembrolizumab, Chemotherapy, Radiation, Surgery)
Number analyzed (Participants) | 31
percentage of patients | 22.6 [11.4 to 39.8]

2. Secondary Outcome: Complete Resection With no Tumor Within 1 mm of the Resection Margins (R0) Rate
Description: Defined as the number of patients who achieve R0 resection divided by total number of evaluable patients.
Time Frame: Up to 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Pembrolizumab, Chemotherapy, Radiation, Surgery)
Number analyzed (Participants) | 31
Participants | 28

3. Secondary Outcome: Disease-free Survival (DFS)
Description: Defined as the time from the date of study registration to the date of death due to any cause
Time Frame: Up to 3 years
Population: All patients that achieved an R0
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Pembrolizumab, Chemotherapy, Radiation, Surgery)
Number analyzed (Participants) | 27
months | 8.87 [7.46 to NA] — Upper limit on 95% confidence interval is not estimable (NE), due to an insufficient number of participants with events.

4. Secondary Outcome: Time to Relapse (TTR)
Description: Defined as the time from the date of study registration to the date of 1st documented relapse/recurrence among patients who achieve R0 resection
Time Frame: Up to 3 years
Population: All patients that achieved an R0
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Pembrolizumab, Chemotherapy, Radiation, Surgery)
Number analyzed (Participants) | 27
months | 8.87 [7.46 to NA] — Upper limit on 95% confidence interval is not estimable (NE), due to an insufficient number of participants with events.

5. Secondary Outcome: Overall Survival (OS) at Two Years
Description: The distribution of OS will be estimated using the method of Kaplan-Meier. Two-year OS rate and confidence interval will be estimated based on Kaplan-Meier curve.
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Pembrolizumab, Chemotherapy, Radiation, Surgery)
Number analyzed (Participants) | 31
percentage of participants | 63.3 [47.4 to 84.4]

6. Secondary Outcome: Progression-free Survival (PFS) Rate at Two Years
Description: The distribution of PFS will be estimated using the method of Kaplan-Meier. Two-year PFS rate and confidence interval will be estimated based on Kaplan-Meier curve.
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Pembrolizumab, Chemotherapy, Radiation, Surgery)
Number analyzed (Participants) | 31
percentage of participants | 16.7 [6.0 to 46.5]

7. Secondary Outcome: Number of Patients Experiencing Dose-limiting Toxicities (DLTs)
Description: Assessed by Common Terminology Criteria for Adverse Events (CTCAE) version 4.0. The maximum grade for each type of adverse events that are possibly, probably or definitely related to study treatments will be recorded for each patient.
Time Frame: Up to 3 years
Population: The 16 eligible patients enrolled in the phase 1b portion of the study were assessed for DLTs.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Pembrolizumab, Chemotherapy, Radiation, Surgery)
Number analyzed (Participants) | 16
Participants | 2

ADVERSE EVENTS:
Time Frame: 3 years, 6 months
Arm/Group | Treatment (Pembrolizumab, Chemotherapy, Radiation, Surgery)
All-Cause Mortality (participants affected / at risk) | 11/31
Serious Adverse Events (participants affected / at risk) | 13/31
Other Adverse Events (participants affected / at risk) | 31/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Pembrolizumab, Chemotherapy, Radiation, Surgery) (N=31)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Hemolysis (Blood and lymphatic system disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Pericarditis (Cardiac disorders) | 1 (2)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Endocrine disorders - Other, specify (Endocrine disorders) | 1 (1)
Eye disorders - Other, specify (Eye disorders) | 1 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (2)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 1 (1)
Gastric hemorrhage (Gastrointestinal disorders) | 1 (1)
Gastric perforation (Gastrointestinal disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (2)
Enterocolitis infectious (Infections and infestations) | 1 (1)
Infections and infestations - Oth spec (Infections and infestations) | 2 (2)
Sepsis (Infections and infestations) | 3 (4)
Esophageal anastomotic leak (Injury, poisoning and procedural complications) | 1 (1)
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Investigations - Other, specify (Investigations) | 2 (2)
Lymphocyte count decreased (Investigations) | 2 (2)
Platelet count decreased (Investigations) | 1 (1)
White blood cell decreased (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Resp, thoracic, mediastinal - Oth spec (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Pembrolizumab, Chemotherapy, Radiation, Surgery) (N=31)
Anemia (Blood and lymphatic system disorders) | 8 (11)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Myocarditis (Cardiac disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 2 (2)
Hyperthyroidism (Endocrine disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (2)
Constipation (Gastrointestinal disorders) | 20 (28)
Diarrhea (Gastrointestinal disorders) | 18 (52)
Dysphagia (Gastrointestinal disorders) | 6 (7)
Gastric fistula (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders - Oth spec (Gastrointestinal disorders) | 4 (7)
Ileus (Gastrointestinal disorders) | 2 (2)
Mucositis oral (Gastrointestinal disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 26 (53)
Obstruction gastric (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 14 (30)
Fatigue (General disorders) | 29 (166)
Gen disord and admin site conds-Oth spec (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Allergic reaction (Immune system disorders) | 1 (1)
Abdominal infection (Infections and infestations) | 1 (1)
Pelvic infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Esophageal anastomotic leak (Injury, poisoning and procedural complications) | 2 (2)
Inj, pois and proced complic - Oth spec (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 4 (5)
Alkaline phosphatase increased (Investigations) | 5 (6)
Aspartate aminotransferase increased (Investigations) | 4 (6)
Cardiac troponin I increased (Investigations) | 1 (1)
Cardiac troponin T increased (Investigations) | 1 (1)
Creatinine increased (Investigations) | 6 (8)
Investigations - Other, specify (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 25 (67)
Neutrophil count decreased (Investigations) | 16 (17)
Platelet count decreased (Investigations) | 16 (24)
Weight loss (Investigations) | 3 (7)
White blood cell decreased (Investigations) | 15 (18)
Anorexia (Metabolism and nutrition disorders) | 6 (7)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (3)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Neoplasms benign, mal, uncpec - Oth spec (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 1 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 11 (36)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 11 (25)
Hypertension (Vascular disorders) | 6 (11)
Hypotension (Vascular disorders) | 2 (2)
Thromboembolic event (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-01-28): https://cdn.clinicaltrials.gov/large-docs/46/NCT02730546/Prot_SAP_000.pdf
  • Informed Consent Form (2021-04-23): https://cdn.clinicaltrials.gov/large-docs/46/NCT02730546/ICF_001.pdf